CLINICAL TRIAL: NCT04974294
Title: A Phase IV Double Blind Randomised Controlled Trial (DBRCT) to Investigate the Effect of PCV-13 and PPV-23 on Pneumococcal Colonisation Using the Experimental Human Pneumococcal Challenge (EHPC) Model in Healthy Adults
Brief Title: PREVENTING PNEUMOcoccal Disease Through Vaccination (Study 2)
Acronym: Pneumo 2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19-104
Record Dates: First submitted 2021-07-21; First posted 2021-07-23 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Streptococcus Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — Pneumococcal Vaccines; Heptavalent Pneumococcal Conjugate Vaccine; Sodium Chloride; Injections

STUDY DESIGN:
Intervention Model Description: double blind RCT
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will remain blinded until the completion of the last participant, last study visit (Day 23: 7-month challenge). As the appearance of the vaccines are different, physical blindfolds may be worn by the participant to maintain blinding. This method of blinding has been used by our team previously and the time wearing the blindfold is kept to an absolute minimum for participant comfort. Un-blinded clinical team members will prepare and administer the vaccines/placebo to the participants in a blinded manner, shielding the vaccine formula, syringe and box from the participant when it is administered. The vaccine will be checked and prepared in a separate room to the participant and in a separate location to the blinded team. The participant will be seated in the vaccination room, the un-blinded clinical members will enter the vaccination room immediately prior to administration. Local SOPs will be followed to ensure appropriate participant team blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- PPV23 (Active Comparator)
  Interventions: Biological: PPV23
- PCV13 (Active Comparator)
  Interventions: Biological: PCV13
- Saline placebo (Placebo Comparator)
  Interventions: Other: Saline for injection

INTERVENTIONS:
Biological: PPV23 — random allocation 1:1:1 IM injection
  Other Names: pneumovax
  Arms: PPV23
Biological: PCV13 — random allocation 1:1:1 IM injection
  Other Names: prevenar
  Arms: PCV13
Other: Saline for injection — random allocation 1:1:1 IM injection
  Arms: Saline placebo

SUMMARY:
To determine the effect of PCV-13 and PPV-23 vaccination versus control on experimental pneumococcal colonisation of 2 clades of serotypes 3 and 6B at 1 month and 6 months post vaccination respectively, using the EHPC model.

DETAILED DESCRIPTION:
Streptococcus pneumoniae (SPN) is the leading cause of morbidity and mortality worldwide, causing community acquired pneumonia (CAP), bacterial meningitis and bacteremia. Pneumococcal infections cause over 1 million pneumonia deaths per year in children in the developing world and is a major burden of otitis media globally.

The LSTM Experimental Human Pneumococcal Challenge (EHPC) model is a unique method of measuring pneumococcal colonization of bacteria, understanding the effect of pneumococcal colonization on acquired immunity, and allows vaccines to be tested in adults to understand their effect on colonization in a manner which is cost-effective and uses much smaller numbers of participants compared to large phase III clinical trials.

Participants: Healthy adults aged 18-50 years of age (inclusive) will be recruited. A recruitment target of up to 516 participants with an approximate screen failure/dropout rate of 20% will ensure 410 participants complete Part A and 246 complete Part A & B of the trial.

Methods: Double blind randomized controlled trial (DBRCT) to investigate the effect of PCV-13 and PPV-23 vaccination on pneumococcal colonisation using the EHPC model in healthy adults. Participants will be randomised to 5 arms for Part A of the study that:

1. to receive PCV-13 vaccine IM and inoculation a month later with SPN3 clade 1a;
2. to receive PCV-13 vaccine IM and inoculation a month later with SPN3 clade 2;
3. to receive PPV-23 vaccine IM and inoculation a month later with SPN3 clade 1a;
4. to receive 0.9% saline for injection IM and inoculation a month later with SPN3 clade 1a or
5. to receive 0.9% saline for injection IM and inoculation a month later with SPN3 clade 2.

The last two 0.9% saline of injection groups represent the placebo control groups. The SPN3 (2 clades) is amoxicillin-susceptible. After challenge (inoculation) they will be followed up for 23 days where nasal, blood and urine samples will be taken. Part B of the trial will run 6 months post vaccination. Participants will be re-screened for safety prior to Part B to ensure they remain eligible. The 3 groups of participants detailed below from the Part A population will proceed to Part B of the trial:

1. Up to 104 of the participants that received PCV-13 in Part A (split across clades 1a and 2)
2. Up to 104 of the participants that received PPV-23 in Part A
3. Up to 104 of the participants that received 0.9% saline for injection in Part A (split across clades 1a and 2) The total number to proceed to Part B will be up to 312 to allow for 20% dropout / screen failure to ensure 246 complete part A & B. All Part B Participants will receive a second inoculation of amoxicillin-susceptible SPN6B at 6 months post-vaccine and will be followed up for 23 days in total where further samples will be taken (Trial Flow Chart and Table 2). All participants will take a 5-day course of amoxicillin three times a day (TDS) at the end of Part A to ensure experimental colonization clearance prior to Part B inoculation. Participants that are experimentally colonized at any point following the SPN6B challenge at 6 months (Part B) will take a 3-day course of amoxicillin TDS.

Randomization & Blinding: Participants will be randomized to receive PCV-13 vaccine and clade 1a (group 1), PCV-13 and clade 2 (group 2), PPV-23 vaccine and clade 1a (group 3), 0.9% saline for injection and clade 1a (group 4) or 0.9% saline for injection and clade 2 (group 5) vaccine in a ratio of 1:1:1:1:1 with up to 104 participants in each arm. Randomization will be computer-generated.

Randomization will occur in two cohorts:

1. Cohort I: 312 subjects for five groups 1:1:2:1:1 in block sizes of 6
2. Cohort II: 204 participants for four groups 1:1:0:1:1 in block sizes of 4 This will ensure that overall the randomization ratio is 1:1:1:1:1, but it will allow 312 participants from Cohort I, split equally across participants that have received PCV-13, PPV-23 and placebo to proceed to part B of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-50 years (inclusive)
* Fluent spoken English - to ensure a comprehensive understanding of the research project and their proposed involvement
* Capacity to provide written informed consent
* Females of childbearing potential with a negative urine pregnancy test at screening and willing to practice adequate birth control measures during the study.

Exclusion Criteria:

* Be currently involved in another study unless observational or non-interventional. Exceptions are the EHPC bronchoscopy study and COVID-19 observational and interventional trials. The exceptions will be applied at the discretion of the Chief Investigator to ensure no harm comes to the participants (e.g. excessive blood sampling)
* Be a participant in a previous EHPC trial within the last 3 years (at the discretion of the study team).

  * Vaccination (self-reported or confirmed from GP questionnaire [GPQ] or medical summary if deemed necessary at clinician discretion): Have had any previous pneumococcal vaccination (including in a research study).
  * Allergy:
* Have allergy to penicillin or amoxicillin.
* Have previous anaphylaxis or severe adverse reaction to any component/excipient of the vaccines or to any vaccine.

  • Health history (self-reported by the participant or confirmed in GPQ or medical summary if deemed necessary at clinician discretion): Ill health including but not limited to:
* Asplenia or dysfunction of the spleen.
* Chronic respiratory disease (e.g. asthma [on medication], COPD, emphysema, bronchiectasis).
* Chronic heart disease (e.g. angina, ischaemic heart disease, chronic heart failure) [controlled stable hypertension may be included].
* Chronic kidney disease (e.g. nephrotic syndrome, kidney transplant, on dialysis).
* Chronic liver disease (e.g. cirrhosis, biliary atresia, hepatitis).
* Chronic neurological conditions
* Connective tissue disease
* Dementia
* Diabetes mellitus (including diet controlled).
* Immunosuppression or history of receiving immunosuppressive therapy.
* Individuals with cochlear implants.
* Individuals with major cerebrospinal fluid leaks (e.g. following trauma, major skull surgery, or requiring CSF shunt).
* Recurrent otitis media.

  * Have any uncontrolled medical/surgical conditions (such as but not restricted to mental health conditions, epilepsy, narcolepsy or chronic pain) at the discretion of the study doctor.
  * Major pneumococcal illness requiring hospitalisation within the last 10 years
  * Other conditions considered by the clinical team as a concern for participant safety or integrity of the study.
  * Taking medication:
* That may affect the immune system e.g. steroids, inflammation altering (e.g. nasal steroids, Roaccutane) or disease-modifying anti-rheumatoid drugs.
* Long-term use of antibiotics (see also section 6.3 Temporary exclusion criteria).
* Nitroglycerin
* That affects blood clotting (any oral/injectable anticoagulants [except aspirin]).

  * Female participants who are pregnant, lactating or intending on becoming pregnant during the study.
  * Direct caring role or close contact with individuals at higher risk of infection (during the challenge period)
* Children under 5 years age.
* Chronic ill health or immunosuppressed adults.
* People that are part of the extremely vulnerable group as defined by Public Health England (PHE)

  • Smoker:
* Current or ex-smoker (regular cigarettes/cigars/e-cigarette/vaping/smoking of recreational drugs) in the last 6 months.
* Previous significant smoking history (more than 20 cigarettes per day for 20 years or the equivalent [>20 pack years]).

  * History or current drug or alcohol abuse (frequently drinking alcohol): men and women should not regularly drink >3 units/day and >2 units/day respectively) at discretion of the clinician.
  * Significant mental health problems (uncontrolled condition or previous admission in a psychiatric unit, at the discretion of the clinician) that would impair the participant's ability to participate in the study
  * Overseas travel planned: Overseas travel during the follow-up period Part A or Part B.
  * Participants who meet STOP criteria at the time of screening, as detailed in Table 4.
  * Any other issue which, in the opinion of the study staff, may
* Put the participant or their contacts at risk because of participation in the study,
* Adversely affect the interpretation of the study results, or
* Impair the participant's ability to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 516 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of experimental pneumococcal colonisation with SPN3 determined by the presence of pneumococcus in nasal wash (NW) by classical culture or molecular methods | any time point during 23 days following experimental human pneumococcal challenge (EHPC) 1 month after vaccination in the PCV-13, PPV-23 and control groups.
  The rate of experimental pneumococcal colonisation with SPN3 determined by the presence of pneumococcus in nasal wash (NW) by classical culture or molecular methods at any time point during 23 days following experimental human pneumococcal challenge (EHPC) 1 month after vaccination in the PCV-13, PPV-23 and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Liverpool School of Tropical Medicine, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liatsikos K, Hyder-Wright A, Pojar S, Chen T, Wang D, Davies K, Myerscough C, Reine J, Robinson RE, Urban B, Mitsi E, Solorzano C, Gordon SB, Quinn A, Pan K, Anderson AS, Theilacker C, Begier E, Gessner BD, Collins A, Ferreira DM; PNEUMO 2 study group. Protocol for a phase IV double-blind randomised controlled trial to investigate the effect of the 13-valent pneumococcal conjugate vaccine and the 23-valent pneumococcal polysaccharide vaccine on pneumococcal colonisation using the experimental human pneumococcal challenge model in healthy adults (PREVENTING PNEUMO 2). BMJ Open. 2022 Jul 7;12(7):e062109. doi: 10.1136/bmjopen-2022-062109. PMID 35798520